CLINICAL TRIAL: NCT03821168
Title: The Effect of Intravitreal Erythropoietin Injection for Refractive Diabetic Macular Edema
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Zahra Rabbani Khah, Clinical Professor, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 95287
Record Dates: First submitted 2018-12-27; First posted 2019-01-29 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2018-12

CONDITIONS: Refractory Diabetic Macular Edema
MeSH Terms: interventions — Erythropoietin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intravitreal injection of bevacizumab and erythropoietin (Active Comparator): erythropoietin:
  Interventions: Drug: injection of bevacizumab and erythropoietin
- intravitreal injection of bevacizumab (Active Comparator): bevacizumab:1.25 mg
  Interventions: Drug: injection of bevacizumab

INTERVENTIONS:
Drug: injection of bevacizumab and erythropoietin — injection of bevacizumab and erythropoietin
  Arms: intravitreal injection of bevacizumab and erythropoietin
Drug: injection of bevacizumab — under gone 3 intravitreal injection of bevacizumab monthly and examine monthly for Visual acuity and central macular thickness
  Arms: intravitreal injection of bevacizumab

SUMMARY:
after advent of RD photoreceptor degeneration Occurred. This process appears as a incredible and progressive event that will not stop till reattachment of RPE and neurosensory retina happened .

Process of degeneration begins from first hours of RD establishment Neuroprotection of photoreceptor following RD is a novel and debatable discussion encountered in recent years .

How to stop this phenomena and neuroprotective agent role in this issue are a new interest of researches.

In the study investigators are planning to perform a clinical trial to demonstrate the minocycline neuroprotective effect in a double blind design as this impact has been implicated previously in a animal study.

ELIGIBILITY:
Inclusion Criteria:

* Patient with refractory diabetic macular edema at least one month after third injection

Exclusion Criteria:

* previous vitreoretinal surgery previous glaucoma surgery glaucomatous patient open heart surgery active proliferative diabetic retinopathy one eye patients vitreous hemorrhage

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2019-03-01 (Estimated); Primary Completion 2019-04-01 (Estimated); Study Completion 2019-10-01 (Estimated)

PRIMARY OUTCOMES:
best corrected visual acuity | 1 month
  Snellen chart

SECONDARY OUTCOMES:
Optical coherence tomography | 1 month
  Optical coherence tomography

CONTACTS AND LOCATIONS:
Locations (1):
- Ophthalmic Research Center, Tehran, Iran

REFERENCES:
- [Derived] Entezari M, Flavarjani ZK, Ramezani A, Nikkhah H, Karimi S, Moghadam HF, Daftarian N, Yaseri M. Combination of intravitreal bevacizumab and erythropoietin versus intravitreal bevacizumab alone for refractory diabetic macular edema: a randomized double-blind clinical trial. Graefes Arch Clin Exp Ophthalmol. 2019 Nov;257(11):2375-2380. doi: 10.1007/s00417-019-04383-2. Epub 2019 Aug 10. PMID 31401683